CLINICAL TRIAL: NCT07048392
Title: Retrieval-Based Word Learning in Developmental Language Disorder During Book Reading II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laurence Leonard, Professor, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1603017480E; R01DC014708 (NIH)
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Developmental Language Disorder and Language Impairment; Specific Language Impairment; Language Development
Keywords: word learning; word retrieval; preschool-aged children
MeSH Terms: conditions — Language Development Disorders; Language Disorders; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: Within-participant design in which each child learns words under two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Developmental Language Disorder (Experimental): These children have a significant delay in language development in the absence of hearing impairment, cognitive delay, autism, or neurological injury/disease.
  Interventions: Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based word learning: Repeated Study condition
- Children with typical language development (Experimental): Children whose language development is as expected for their age.
  Interventions: Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based word learning: Repeated Study condition

INTERVENTIONS:
Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition — Each child will learn 8 novel nouns referring to unfamiliar plants and animals ("nepp") and a related "meaning" ("a nepp likes rain") in the context of a story book. Four of the nouns will be will be learned using repeated spaced retrieval. In this condition, they will initially hear the information and be asked to retrieve it. Thereafter, they will be asked to retrieve it after hearing 3 intervening words. After each retrieval attempt, they will hear the target information again. This procedure will occur on two consecutive days.
Behavioral: Retrieval-based word learning: Repeated Study condition — Each child will learn 8 novel nouns referring to unfamiliar plants and animals ("nepp") and a related "meaning" ("a nepp likes rain") in the context of a story book. Four of the nouns will be will be learned using repeated study trials only (with no retrieval practice). In this condition, they will simply hear the information (word & meaning) as part of the story. This procedure will occur on two consecutive days.

SUMMARY:
Children with developmental language disorder (DLD; also referred to as specific language impairment) experience a significant deficit in language ability that is longstanding and harmful to the children's academic, social, and eventual economic well-being. Word learning is one of the principal weaknesses in these children. This project focuses on the word learning abilities of four- and five-year-old children with DLD. The goal of the project is to build on the investigators' previous work to determine whether, as has been found thus far, special benefits accrue when these children must frequently recall newly introduced words during the course of learning. In this study, the investigators seek to replicate the advantage that repeated retrieval holds over simple exposure to the words appearing in the context of a story book by increasing the degree to which the words are integrated into the story line.

DETAILED DESCRIPTION:
Developmental Language Disorder (DLD) affects language learning in an estimated 7% of children. Although much of the research literature has emphasized difficulties learning grammar, children with DLD also have major deficits in vocabulary. In recent work, the investigators have been examining the benefit of retrieval practice to enhance word learning and retention in preschoolers with DLD. The rationale behind this work is grounded in the growing literature in the field of cognitive psychology which shows that repeated practice in retrieving information results in greater long-term retention than continuous study of that information without opportunities for retrieval. In addition, retrieval practice that occurs after a delay-or "spacing" between study of a word and subsequent recall attempts-can lead to stronger effects.

The investigators have explored the benefits of retrieval practice for preschoolers with DLD and with typical language development (TD), showing that recall and retention for novel words (nouns, adjectives, verbs) were greater when learned using repeated spaced retrieval (RSR) than when learned using repeated study only. Despite benefiting from RSR, children with DLD still showed lower levels of recall than children with TD.

In the investigators' immediately preceding study, the same words and retrieval schedules used in earlier studies were embedded into story contexts. Artist-illustrated stories incorporated illustrations of the unfamiliar plants and animals that served as referents of novel nouns. The findings of greater learning with RSR than with RS were replicated. However, in that study, the words were merely mentioned in the story, as objects that the characters happened to see along their journey. In this new study, the words to be learned are more tightly integrated into the story line, to more closely approximate the everyday shared book reading that occurs in homes, preschools, and clinics. Sixteen children with DLD will be recruited for this study along with 16 children with TD matched on chronological age. Using a within-subjects design, children will learn eight novel nouns, four embedded in each story. Along with each word form, children will learn a "meaning", that is, an additional piece of semantic information about the referent.

For words in the RSR condition, each novel word and meaning, paired with its referent, will be presented as part of the story. Immediately after hearing it, children will be asked to recall both form and meaning, and then will hear those repeated. All subsequent retrieval trials will occur after three other words have intervened since the last time the word appeared in a study trial. Novel words assigned to the comparison condition will simply be heard paired with their referent during the story at the same frequency as words in the RSR condition. Children will not be asked to recall the words in the comparison condition during the learning period. Stories will be presented twice, on two consecutive days. As written, children will hear the words the same number of times overall as in the investigator's previous studies, allowing evaluation of the benefits of the story format. Recall of the word forms and meanings will be tested after the story book reading on both the first and second days. One week later, the recall test will be re-administered and children will complete a three-alternative recognition test.

The investigators hypothesize that the findings will replicate the findings of their immediately preceding study, this time with the words integrated to a greater extent within the stories, thus more closely approximating the more typical shared book reading experienced by children. Specifically, the children will show greater recall for word forms and meanings in the RSR condition than those in the repeated study condition. Past studies have not consistently shown an advantage for recognition; therefore, we do not predict a difference for this particular measure. It is also expected that children with TD will remember more words overall than children with DLD. To the degree that the story format is more engaging for children, overall recall will be enhanced for both groups. Assuming that the results are replicated, it is hoped that the children's book reading format will prove amenable for use by teachers and speech-language pathologists who work with children with DLD.

ELIGIBILITY:
Inclusion Criteria:

* a significant deficit in language ability (language test score below cutoff for best sensitivity/specificity) or documented age-appropriate language ability.
* normal hearing.
* no evidence of neurological damage or disease.
* scores on tests of nonverbal intelligence above the intellectual disability range
* not within Autistic range on Autism screening test
* native English speaker (can be bilingual)

Exclusion Criteria:

* failed hearing screening
* known neurological damage or disease
* scores on tests of nonverbal intelligence below the intellectual disability range (standard score less than 75)
* autism spectrum disorder
* non-native English speaker

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Word Form Recall Accuracy (number of words correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, Day 1 | 5 minutes after end of first (Day 1) learning period
  Child is asked to recall and say the word associated with each novel referent.
Word Form Recall Accuracy (number of words correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, Day 2 | 5 minutes after end of first (Day 2) learning period
  Child is asked to recall and say the word associated with each novel referent.
Word Form Recall Accuracy (number of words correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, One week | One week after end of learning period
  Child is asked to recall and say the word associated with each novel referent.
Word Meaning Recall Accuracy (number of semantic associations correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, Day 1 | 5 minutes after end of first (Day 1) learning period
  Child is asked to recall and say semantic information associated with the novel referent.
Word Meaning Recall Accuracy (number of semantic associations correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, Day 2 | 5 minutes after end of first (Day 2) learning period
  Child is asked to recall and say semantic information associated with the novel referent.
Word Meaning Recall Accuracy (number of semantic associations correctly recalled) in Repeated Spaced Retrieval and Repeated Study conditions, one week | One week after end of learning period
  Child is asked to recall and say semantic information associated with the novel referent.
Word recognition (number of words accurately identified) in repeated spaced retrieval and repeated study conditions. | One week after end of learning period
  Upon hearing a novel word, the child is asked to indicate (by pointing) which picture among 4 options is referred to.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence B. Leonard, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that contribute to our final published results will be made available at clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the results are published or within 12 months from the primary completion date (i.e., the date of final data collection for the primary outcome measure).
Access Criteria: De-identified data will be made publicly available at www.clinicaltrials.gov